CLINICAL TRIAL: NCT01947296
Title: Evaluation of the Impact of a Coordinated Regional Organization to Secure Patient's Care Treated by Oral Antineoplastic Agents
Brief Title: Impact of a Coordinated Regional Organization to Secure Patient's Care Treated by Oral Antineoplastic Agents
Acronym: CHIMORAL
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: oncorif (Unknown)
Responsible Party: Sponsor
Other Study IDs: NI 12019; C1204 (Other: ANSM)
Record Dates: First submitted 2013-09-02; First posted 2013-09-20 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Cancer
Keywords: Oral antineoplastic agent; Adverse Effects; Cancer Networks; Continuity of care; Coordination of patient's care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group " coordinated care": Patient living in place covered by cancer network participating to the study is in the group "coordinated care"
- Group " usual care ": Patient living in place covered by cancer network non participating to the study or without cancer network is in the group "usual care"

SUMMARY:
The purpose is to estimate evolution of patients treated by oral neoplastic agents, in term of early or unforeseen recourse to the hospital for adverse events.

DETAILED DESCRIPTION:
Introduction :

Oral antineoplastic agents know a full development in particular targeted therapies. Their adverse events (AE) lately detected can lead to non compliance or treatment discontinuation which can be at the origin of disease progression. They can also lead to hospitalization or recourse to emergency department associating to cost for the society.

Hypothesis :

A coordinated intervention of cancer network in relation with primary healthcare professionals, would improve safety of care's patient treated with oral antineoplastic agent by preventing serious AEs through rapid detection.

Primary objective :

The primary objective is to estimate the effect of coordinated intervention of cancer network, in terms of number of early or unforeseen recourses to hospital for AE, within the first 6 months after oral neoplastic agent introduction.

Secondary objectives :

The secondary objective is to estimate the effect of coordinated intervention of cancer network, within the first 6 months after oral neoplastic agent introduction, in terms of number of hospitalization for AE, number of consultation for AE, number of early or unforeseen recourses to hospital for grade 1 / 2 AE, number of AE per detection grade, AE maximal grade, AE all grade, disease progression, the global survival (death for any causes and for AE), drug dose-intensity taken by the patient during his treatment, number of recourses to the health care system, quality of life, patient's satisfaction, medical economic evaluation

Primary outcome :

The main outcome is the number of early or unforeseen recourses to hospital for AE.

Secondary outcomes :

The secondary outcomes are all deaths and deaths from AE, number of hospitalization for AE, number of consultation for AE, number of early or unforeseen recourses to hospital for grade 1 / 2 AE, disease progression, drug dose-intensity taken by the patient during his treatment, number of recourses to the health care system, number of AE per detection grade, AE maximal grade, AE all grade, quality of life, patient's satisfaction, medical economic evaluationMethodology, design :

A comparative, controlled, not randomized, multicenter, prospective, "quasi-experimental" study, allows estimating evolution of patients according to the existence of a cancer network in their residence place.

Number of needed subjects: 440 patients.

Total duration of the study: 27 months. Inclusion Period: 21 months. length of participation period for one patient: 6 months. Number of participating centers: 21. Average number of inclusions a month by center: 4.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by cancer (breast, colorectal, liver, lung, kidney, gastrointestinal stromal tumor, pancreas)
* treated by capecitabine, erlotinib, gefitinib, imatinib, lapatinib, sorafenib, sunitinib, vinorelbine, Evérolimus, Pazopanib, Etoposide, Topotécan
* 18 years old or more

Exclusion Criteria:

* refusal to participate
* lack proficiency in French ,
* having a Performance Status > 2,
* home based care,
* patient enrolled in clinical trials
* patient enrolled in therapeutic education program
* patient under administrative supervision or legal guardianship
* not affiliated with Patient Social Security or CMU (recipient or beneficiary)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with oral antineoplastic agent introduction in the region of Ile-de-France
Sampling Method: Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of early or unforeseen recourses to hospital for adverse event. | within the first 6 monts after oral neoplastic agent introduction

SECONDARY OUTCOMES:
all deaths and deaths from AE | within the first 6 monts after oral neoplastic agent introduction
number of hospitalization for AE | within the first 6 monts after oral neoplastic agent introduction
number of consultation for AE | within the first 6 monts after oral neoplastic agent introduction
number of early or unforeseen recourses to hospital for grade 1 / 2 AE | within the first 6 monts after oral neoplastic agent introduction
disease progression | within the first 6 monts after oral neoplastic agent introduction
drug dose-intensity taken by the patient during his treatment | within the first 6 monts after oral neoplastic agent introduction
number of recourses to the health care system | within the first 6 monts after oral neoplastic agent introduction
number of AE per detection grade, AE maximal grade, AE all grade | within the first 6 monts after oral neoplastic agent introduction
quality of life | within the first 6 monts after oral neoplastic agent introduction
patient's satisfaction | within the first 6 monts after oral neoplastic agent introduction
  patient's satisfaction will be characterized with a questionnaire
medical economic evaluation | within the first 6 monts after oral neoplastic agent introduction
  Medical economic evaluation use The incremental cost-effectiveness ratio (ICER. This is an equation used commonly in health economics to provide a practical approach to decision making regarding health interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-¨Pierre Lotz, Professor, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided